CLINICAL TRIAL: NCT04998552
Title: Safety and Efficacy of Cyberknife in Patients With Borderline Resectable or Locally Advanced Pancreatic Adenocarcinoma: Open Label Prospective Randomized Clinical Trial
Brief Title: Safety of Cyberknife in Patients With Borderline Resectable or Locally Advanced Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Health System, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PANCAN SBRT
Record Dates: First submitted 2021-07-20; First posted 2021-08-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Pancreas Adenocarcinoma
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: The study is an open-label, longitudinal, prospective randomized, superiority clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SBRT (Cyberknife) (Experimental): 5-10 Gy/fraction. Average of 45 minutes every other day for a total of 5 sessions (1.5-2 weeks).
  Interventions: Radiation: Cyberknife
- IMRT (Active Comparator): 1.2-3 Gy/fraction up to 40 fractions. 15 mins daily (M-F) for a total of 28 sessions (5.5 weeks).
  Interventions: Radiation: Cyberknife

INTERVENTIONS:
Radiation: Cyberknife — 5-10 Gy/fraction.Average of 45 minutes every other day for a total of 5 sessions (1.5-2 weeks).

SUMMARY:
The hypothesize that SBRT will limit or reverse tumor growth and thereby convert the borderline resectable disease or locally advanced disease in to a resectable tumor. Furthermore, we want to assess whether SBRT leads to an improved quality of life compared to IMRT.

DETAILED DESCRIPTION:
The study is an open-label, longitudinal, prospective randomized, superiority clinical trial. The protocol applies to patients with confirmed diagnosis of pancreatic adenocarcinoma and pancreatic protocol CT scan showing borderline resectable disease or locally advanced disease as per the NCCN guidelines (See addendum, NCCN Guidelines 2021, PANC-3 and PANC-4). All cases will be discussed at the multidisciplinary GI cancer conference (tumor board). Cases will continue to be reviewed at different milestones of their treatment as described below.

Patients diagnosed with borderline resectable or locally advanced pancreatic cancer will receive standard of care and neoadjuvant chemotherapy according to NCCN guidelines and protocols followed by radiation therapy. The radiation therapy will start 4 weeks after ending the chemotherapy, thereby creating a wash-out period. At the start of the radiation therapy subjects will be consented and randomized into either receiving the IMRT protocol or the SBRT protocol. Baseline measurements will be collected at the start of the radiation treatment. At the completion of the radiation therapy the subject's progress and condition will be evaluated by the tumor board and a multidisciplinary consensus agreement will be reached to decide the course of further treatment, which could be chemotherapy (if deemed unresectable) or proceed with surgery (if deemed resectable). Irrespective the decision, patients will be asked to return for follow up every 3 months to obtain CT scans, assess quality of life and provide a biological sample (blood) for up to 12 months after the initiation of the radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Able to sign the informed consent and understand the consenting process
* Completed neoadjuvant chemotherapy regimen
* Patient is 18 years of age and older
* Eastern Cooperative Oncology Group (ECOG) Status of 0-1.
* Patient has a diagnosis of Stage I to Stage III pancreatic cancer cytologically or pathologically confirmed per American Joint Committee on Cancer (AJCC) staging criteria and NCCN guidelines, based on radiographic imaging or exploratory laparoscopic surgery, low degree of arterial involvement (CA, CHA, SMA) and no aorta involvement.
* Patients who are deemed eligible for IMRT or SBRT and approved to receive radiation therapy by multidisciplinary tumor board
* Patient shows no evidence of disease progression to distant metastasis based on NCCN.
* Negative pregnancy test

Exclusion Criteria:

* Pregnant or lactating female patients of reproductive potential who are not willing to employ highly effective birth control from screening to 6 months after the last dose of radiation therapy.
* Resectable pancreatic cancer (See addendum, NCCN Guidelines 2021, PANC-2)
* Unresectable pancreatic cancer (See addendum, NCCN Guidelines 2021, PANC-6)
* Patients who are unable to tolerate general anesthetic with full skeletal muscle blockade.
* Patients with implanted cardiac pacemakers, defibrillators, electronic devices or implanted devices with metal parts in the thoracic cavity.
* Life expectancy of < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2027-06-22 (Estimated); Study Completion 2027-06-22 (Estimated)

PRIMARY OUTCOMES:
Resectability | 1 month after the completion of radiation therapy.
  Occurrence of meeting resectability criteria using NCCN (PAN-C) guidelines

SECONDARY OUTCOMES:
Patient Reported Outcome (General) - European Organization for Research and Treatment of Cancer (EORTC). | at baseline and then at 3 month intervals.
  Change in mean score from baseline of Quality of Life using EORTC QLQ-C30 questionnaire. Raw score is transformed to standardize with a lowest value of 0 and a highest of 100.
Patient Reported Outcome (Specific)European Organization for Research and Treatment of Cancer (EORTC). | At baseline and then at 3 month intervals.
  Change in mean score from baseline of Quality of Life using EORTC PAN26 questionnaire. Raw score is transformed to standardize with a lowest value of 0 and a highest of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Shirnett Williamson, MD, Principal Investigator — Capital Health System, Inc
Locations (1):
- Capital Health Medical Center-Hopewell, Pennington, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No